CLINICAL TRIAL: NCT05835375
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy of EQ-778 on Upper Respiratory Tract Health Status in Healthy Adults
Brief Title: A Study to Evaluate the Efficacy of EQ-778 on Upper Respiratory Tract Health Status in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PL/221201/EQ/CCI
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EQ-778 (Active Comparator): 1. capsule to be taken daily after breakfast (in case no URTI episode)
  2. capsules to be taken daily after breakfast (in case of URTI episode)
  Interventions: Other: EQ-778
- Placebo (Placebo Comparator): 1. capsule to be taken daily after breakfast (in case no URTI episode)
  2. capsules to be taken daily after breakfast (in case of URTI episode)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: EQ-778 — 1. capsule daily after breakfast (in case of no URTI episode);
  2. capsules after breakfast (in case of URTI episode)
  Arms: EQ-778
Other: Placebo — 1. capsule daily after breakfast (in case of no URTI episode);
  2. capsules after breakfast (in case of URTI episode)
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, Placebo Controlled study to evaluate the efficacy of 180 days administration of EQ-778 on upper respiratory tract health status in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals ≥ 18 and ≤ 50 years' old with moderate physical activity level as per International Physical Activity Questionnaire - Short Form (IPAQ - SF)
2. BMI ≥ 18.5 and ≤ 34.9 kg/m2
3. High susceptibility to URTIs (≥ 3 and ≤ 6 episodes within 12 months)
4. Commitment to adhere to routine diet and physical activity.
5. Willing to consume IP or placebo, complete questionnaires, records, etc., associated with the study and to complete all clinical study visits.

Exclusion Criteria:

1. History of rhinitis medicamentosa, anatomical nasal obstruction or deformity, nasal reconstructive surgery, etc.
2. Known sensitivity to the investigational product or any excipients of the drug product.
3. Any clinically significant abnormalities of the upper respiratory tract (such as stridor, laryngomalacia, etc)
4. Any clinically significant acute or chronic respiratory illness (such as Sinusitis, pharyngitis/tonsillitis, etc)
5. Chronic cough of any origin
6. Any individual not willing to follow the abstinence from any home-based remedies for common cold such as steam inhalation, decoctions, vapour rub, etc.
7. Individuals with uncontrolled type 2 diabetes as assessed by fasting blood glucose ≥ 126 mg/dL
8. Individuals with uncontrolled hypertension on medication and with systolic blood pressure ≥160 and/or diastolic blood pressure ≥100 mm Hg will be excluded.
9. Unable to abstain from herbal or dietary supplements for URTI throughout the study period.
10. Vaccination against influenza or swine flu within 3 months prior to screening.
11. Individuals with COVID infection in the last 30 days
12. Those who have taken or should be taking or are taking antibiotics, antivirals, steroids, nasal decongestants, antihistamines, NSAIDS (paracetamol) or other medications that are expected to alleviate cold symptoms within two weeks prior to screening.
13. History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.
14. Participation in other clinical trials in last 30 days prior to screening
15. Individuals with substance abuse problems (within 2 years) defined as:

    1. Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine, tobacco or smoking dependence.
    2. High-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week for women and 5 or more alcohol containing beverages on any day or 15 or more alcohol containing beverages per week for men.
16. Individuals who have clinically significant following severe illness (i.e., Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, gastrointestinal diseases, etc.)
17. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
18. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 374 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-04-26 (Estimated); Study Completion 2024-04-26 (Estimated)

PRIMARY OUTCOMES:
To assess effect of administration of IP on the severity of Upper respiratory tract infections (URTI) symptoms as assessed by area under curve (AUC) for Wisconsin Upper Respiratory Symptom Survey - 21 (WURSS-21) symptom severity score. | 180 Days

SECONDARY OUTCOMES:
To evaluate the effect of the IP as compared to placebo | During episodes of URTI throughout the study
  Nasal Viral load as assessed by TRU-PCR analysis
To evaluate the effect of the IP as compared to placebo | On every visit (Day 0, Day 30, Day 60, Day 90, Day 120, Day 150, and Day 180)
  Change in participants' URTI symptoms severity as compared to the previous day
To evaluate the effect of the IP as compared to placebo | On every visit (Day 0, Day 30, Day 60, Day 90, Day 120, Day 150, and Day 180)
  Change in frequency of current URTI episodes rates as compared to the self-reported historical frequency of URTI in previous 6 months before study begins
To evaluate the effect of the IP as compared to placebo | On every visit (Day 0, Day 30, Day 60, Day 90, Day 120, Day 150, and Day 180)
  Percentage of population suffering having one or more episode of URTIs during study.
To evaluate the effect of the IP as compared to placebo | On every visit (Day 0, Day 30, Day 60, Day 90, Day 120, Day 150, and Day 180)
  The time taken for resolution of the symptoms of the URTIs by eDiary records
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150, and Day 180
  Change in quality of life using the WURSS-21 questionnaire (in eDiary, as and when the subject gets an episode - recall period: last 24 hours)
To evaluate the effect of the IP as compared to placebo | Day 0 and Day 180
  Immunity as assessed by the change in salivary IgA from baseline
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150 and Day 180
  Sleep quality assessed by Pittsburgh Sleep Quality Index
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150 and Day 180
  Mood as assessed by Visual Analogue Scale (VAS)
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150, Day 180 and during each URTI episode
  Stress measured by Perceived Stress Scale (PSS)
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150 and Day 180
  General fatigue as assessed by Fatigue Severity Scale (FSS)
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150 and Day 180
  To assess the effect of the IP on the consumption of rescue medication
To evaluate the effect of the IP as compared to placebo | Day 0, Day 30, Day 60, Day 90, Day 120, Day 150 and Day 180
  To assess the impact of the intervention on daily routine activities by a VAS scale
To evaluate the effect of the IP as compared to placebo | On the last day of the URTI episode.
  To assess the impact of the IP on mood, stress, fatigue, sleep quality and physical activity as assessed by a VAS scale

CONTACTS AND LOCATIONS:
Locations (13):
- India (13):
  - V S General Hospital, 239, E-Ward, 2nd floor, Trauma Centre, VS General Hospital, Paldi, Ahmedabad, Gujarat
  - Poojan Multispeciality Hospital, Navnidhi Avenue, Shubhash Chowk, Swami Vivekanand Marg, Near, Memnagar, Ahmedabad, Gujarat
  - AIMS Hospital, M.I.D.C., Rd Number 5, Milap Nagar, Dombivli East, Dombivali, Maharashtra
  - Shreepad ENT and Head and Neck Hospital, T-3-5, Third Floor, Hare Krishna Plaza Building, Hirawadi Corner, Opp Panchavati Bus Depo, Nashik, Maharashtra
  - Dr. Desale's Joint Clinic, 1st Floor, Canada Complex, Above Sagar Sweet, College Road, Nashik, Maharashtra
  - Life Care Hospital, Life Care Hospital, Mumbai-Agra Highway, Lekha Nagar, Nashik, Maharashtra
  - Dhanwantri Hospital, Pune, Maharashtra
  - Umarji Mother and Child Care Hospital, Balewadi Phata, Baner, Pune, Maharashtra
  - Shatayu, Multispeciality Hospital, Sr no. 275/1, Times Square Building, Bhatewara Nagar, Hinjawadi, Pune, Maharashtra
  - Gayatri Hospital, 16, 17, 18, Lavdeep Building, Waliv, Vasai East, Vasai, Maharashtra
  - Care n Cure Multispeciality Hospital, Kamdhenu Society, Achole Road, Nallasopara East, Virār, Maharashtra
  - Janta Hospital & Maternity Centre, Varanasi, Uttar Pradesh
  - Tulsi Hospital, Delhi